CLINICAL TRIAL: NCT06522022
Title: Comparing Two Screening Approaches for PTSD to Improve Health Outcomes in Pregnant Black Women
Brief Title: PTSD Screening in Pregnant Black Women
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other); University of Missouri, Kansas City (Other)
Responsible Party: Principal Investigator, Abigail Lott, Associate Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00007909
Record Dates: First submitted 2024-07-22; First posted 2024-07-26 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Pregnancy Early; PTSD
Keywords: Pregnancy; Black Women; Screening for Maternal PTSD; Obstetric Care; African-American Women
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Culturally Responsive SBIRT for OB (Experimental): Participants randomized to Culturally Responsive SBIRT for OB will participate in the intervention visit (20-30 minutes) while waiting for their OB visit (or after the visit if time does not allow) and then engage in their prenatal care visit as usual. If any safety concerns emerge during the visit, the lay provider will contact the clinical staff on the study
  Interventions: Behavioral: Culturally Responsive SBIRT for OB
- Brief Screening for PTSD (Experimental): Participants randomized to Brief Screening For PTSD, screening will be conducted as part of regular clinic activities during the initial prenatal care visit. Specifically, clinic staff (nurse, PA) or study staff will ask the questions in the PC-PTSD-5 along with the standard procedure to administer the Edinburgh Postnatal Depression Scale (EPDS), and the provider will review the results with the patient during the prenatal care visit and provide referral resources regardless of screen outcome. Positive PTSD screens (PC-PTSD-5 ≥ 3) will be referred to the hospital's integrated care team following the same model as positive EPDS screens.
  Interventions: Behavioral: Brief Screening for PTSD

INTERVENTIONS:
Behavioral: Culturally Responsive SBIRT for OB — SBIRT is a well-established enhanced screening preventive intervention model that is feasible and acceptable for use with trauma-exposed patients and in minoritized communities and can be delivered in the OB clinic during a prenatal care visit. The elements include:
  1. standardized screening for PTSD and depression using the Primary Care Post Traumatic Stress Disorder Screen (PC-PTSD-5) and the Edinburgh Postnatal Depression Screening (EPDS) that will mirror brief screening practice;
  2. explicit focus on concerns regarding mistrust,
  3. psychoeducation on PTSD, depression, and the effects of trauma including medical trauma and traumatic loss on health/functioning,
  4. motivational interviewing strategy components to promote awareness of psychological symptoms and engagement in culturally relevant resources including support/resources related to relevant social determinants of health,
  5. teaching coping skills with culturally responsive technology tools
  Other Names: Screening Preventive Intervention Model
  Arms: Culturally Responsive SBIRT for OB
Behavioral: Brief Screening for PTSD — This well-established 5-minute in-clinic interview includes administration of the PC-PTSD-5, a 5-item PTSD screening tool by trained medical staff (nurse, physician's assistant). Providers receive approximately one hour of training in trauma-informed care and how to administer the screening protocol. This method is regularly used in primary care clinic settings with trauma-exposed veterans and is validated for use in civilian samples, including low-income Black adults utilizing urban safety net hospital medical clinics.
  Other Names: Standard Screening
  Arms: Brief Screening for PTSD

SUMMARY:
This study will compare the effectiveness of two active screening interventions in improving post-traumatic stress disorder (PTSD) symptoms, maternal perinatal care utilization, satisfaction utilization of mental healthcare services, and maternal health and birth-related outcomes for Black pregnant women.

DETAILED DESCRIPTION:
Researchers will examine whether Culturally Responsive Screening, Brief Intervention, and Referral to Treatment (SBIRT) for obstetrics (OB) is more effective in reducing PTSD symptoms compared to brief screening for PTSD. This study will help participating OB clinics to determine the best option for screening for PTSD in Black pregnant persons in their clinic during first-trimester prenatal visits.

The study population will include Black pregnant women receiving medical care in their first trimester of pregnancy. Surveys and chart abstraction will be used in this study to collect data. The approximate study duration for individuals is 4 visits over 12 months.

ELIGIBILITY:
Inclusion Criteria:

* 18+ years old,
* Ability to provide informed consent,
* English-speaking,
* Willingness to participate in the study,
* Self-identification as Black or African American,
* Pregnant and in the first trimester attending initial prenatal care visit,
* Endorsement of at least one traumatic event in their lifetime.

Exclusion Criteria:

* Active suicidality

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnant Females in their first trimester
Enrollment: 804 (Estimated)
Dates: Start 2025-02-20 (Actual); Primary Completion 2029-03 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
PTSD Checklist for Diagnostic and Statistical Manual of Mental Disorders (DSM)-5 (PCL-5) Score | Initial OB visit (weeks 1-13), second trimester (Weeks 14 to 27), third trimester (weeks 28-40), and 6-weeks postpartum
  Researchers will use the PTSD Checklist for DSM-5 (PCL-5) to measure PTSD symptoms, a well-validated and widely used 21-item measure that assesses the frequency of current PTSD symptoms. Participants report how often they have been bothered by specific symptoms of PTSD on a scale of 0 (not at all) to 4 (extremely). The total symptom severity score ranges from 0 to 80. A provisional PTSD diagnosis can be made and a PCL-5 cut-point score of 33 is recommended.

SECONDARY OUTCOMES:
Adequacy of prenatal care utilization (APNCU) | 6 weeks postpartum
  OB physicians widely use this measure. The APNCU includes what trimester prenatal care began within the index. APNCU is a standard metric, defined as attending at least 80% of prenatal care visits, adjusting for gestational age. Researchers will use chart abstraction to determine the percent attendance of prenatal care adjusting for gestational age at birth.

CONTACTS AND LOCATIONS:
Overall Officials: Abigail Lott, PhD, ABPP, Principal Investigator — Emory University; Briana Woods-Jaeger, PhD, Principal Investigator — Emory University
Locations (2):
- United States (2):
  - Grady Health System, Atlanta, Georgia
  - Truman Medical Center (TMC) system, Kansas City, Missouri

IPD SHARING:
Plan to Share IPD: No